CLINICAL TRIAL: NCT04655924
Title: Artificial Intelligence in Depression - Medication Enhancement: A Randomized, Patient and Rater Blinded, Active-Controlled Trial of a Hybrid-Classic/Machine-Learning Enabled Clinical Decision Aid for Personalized and Individualized Pharmacological Depression Treatment Selection
Brief Title: Artificial Intelligence in Depression - Medication Enhancement
Acronym: AID-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aifred Health (Industry)
Collaborators: McGill University (Other)
Responsible Party: Sponsor-Investigator, Aifred Health, Clinical Trial Manager, Aifred Health Inc.
Organization: Aifred Health Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUSMD 18-04
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: Depression; Treatment Selection; Decision Support; Artificial Intelligence (AI); Machine Learning (ML)
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The Clinical Decision Aid is a digital health platform that collects patient data and provides reports and analyses to clinicians that can assist them in their decision making about treatment selection and management.
Who Masked: Participant, Investigator
Masking Description: Patient and Rater blinded, Physician partially blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Intervention (Experimental): Intervention delivered to patients by digital health platform.
  Interventions: Device: Clinical Decision Support System
- Active Control (Active Comparator): Intervention delivered to patients by digital health platform.
  Interventions: Device: Clinical Decision Support System

INTERVENTIONS:
Device: Clinical Decision Support System — Clinical Decision Support System using Measurement-Based Care and Digital Decision Support Platform

SUMMARY:
This study will determine the safety and potential effectiveness of a digital health platform aimed at improving treatment outcomes for patients with depression by assisting physicians with clinical decision making about depression treatment.

ELIGIBILITY:
Patient Inclusion Criteria:

* diagnosed with major depressive disorder by a physician using DSM-V criteria
* able to provide informed consent
* patients must confirm that they are comfortable being treated for depression by their physician, who may propose a range of treatment options, such as medications or psychotherapies, consistent with best practice guidelines for depression which are included in the application. Physicians will be required, as in usual practice, to explain treatments to patients and patients will be able to give and withdraw consent for treatment in general or for specific treatments as in usual practice.

Patient Exclusion Criteria:

* bipolar disorder of any type
* inability or unwillingness of the individual to give informed consent
* inability to manage patient in an outpatient setting (i.e. imminent suicidality)
* active major depression is not the main condition being treated (i.e. the patient has depressive symptoms in the context of severe substance abuse or a psychotic disorder, but a primary diagnosis of major depressive episode (MDE) cannot be made or would result in inappropriate care).
* inability to use the tool (i.e. patient cannot interface with a mobile phone or computer due to delirium, or another medical condition)* *Note that for patients who do not have access to mobile or desktop devices but are able to use them or to be trained to use them, these will be provided to them at no cost.

Physician Inclusion Criteria:

* any family doctor/primary care physician or psychiatrist accredited in Canada or the USA who treats patients with depression on at least a monthly basis, as well as residents from these specialities supervised by a participating physician
* able to provide informed consent
* comfortable prescribing the range of potential treatments which could have probabilities provided for them by the CDA

No Physician Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Safety - Adverse Events | 3 months
  Adverse and Serious Adverse Events
Effectiveness in Reduction of Depression Symptoms | 3 months
  This is approved as a physician partially-blinded study and, as such, physicians are blinded to the primary outcome.

SECONDARY OUTCOMES:
Time to Remission | 3 months
  To evaluate time to remission between groups. The hypothesis is that time to remission will be shorter in the active intervention group compared to the active control group.
Response Rate | 3 months
  To evaluate response rate between groups. The hypothesis is that the response rate (defined as 50% improvement in symptoms) and time to response, will be higher and lower, respectively, in the active intervention group compared to the active control group.
Patient Disability with WHODAS rating scale | 3 months
  To evaluate between-group differences in patient disability outcomes. The hypothesis is that the physicians in the active intervention arm will produce superior patient outcomes to those physicians using usual guideline-informed practice, in terms of patient function as measured by a rating scale (WHODAS).

OTHER OUTCOMES:
Number of ER visits, admissions, and re-admissions | 3 months
  We will examine impact of health resource utilization by comparing rates of visits, admissions, and re-admissions between groups.
Medication Adherence Rates | 3 months
  We will asses medication adherence rates, as measured by the Brief Adherence Rating Scale, after each visit for the duration of the study and compare between groups.
Patient Questionnaire Response Rate | 3 months
  We will assess the frequency at which patients complete the questionnaires in the digital health platform in both groups.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - VA New Haven, VA Connecticut Healthcare System, West Haven, Connecticut
  - South Florida Veterans Affairs, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Salem VAMC, Salem, Virginia
- Canada (6):
  - CAMH: The Centre for Addiction and Mental Health, Toronto, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - CIUSSS De Centre Ouest De L'île de Montréal, Montreal, Quebec
  - McGill University Health Care Centre (MUHC), Montreal, Quebec
  - CIUSSS De L'Ouest de L'île de Montréal, Montreal, Quebec
  - Douglas Mental Health University Institute, Verdun, Quebec

IPD SHARING:
Plan to Share IPD: Yes
With participating site and on request. Further sharing will be determined at a later date.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: To be determined.

REFERENCES:
- [Derived] Benrimoh D, Whitmore K, Richard M, Golden G, Perlman K, Jalali S, Friesen T, Barkat Y, Mehltretter J, Fratila R, Armstrong C, Israel S, Popescu C, Karp JF, Parikh SV, Golchi S, Moodie EEM, Shen J, Gifuni AJ, Ferrari M, Sapra M, Kloiber S, Pinard GF, Dunlop BW, Looper K, Ranganathan M, Enault M, Beaulieu S, Rej S, Hersson-Edery F, Steiner W, Anacleto A, Qassim S, McGuire-Snieckus R, Margolese HC. Artificial Intelligence in Depression-Medication Enhancement (AID-ME): A Cluster Randomized Trial of a Deep-Learning-Enabled Clinical Decision Support System for Personalized Depression Treatment Selection and Management. J Clin Psychiatry. 2025 Aug 27;86(3):24m15634. doi: 10.4088/JCP.24m15634. PMID 40875536